CLINICAL TRIAL: NCT01620619
Title: The Role of Rotator Interval Closure in Bankart Lesion Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Western Ontario, Canada (Other)
Responsible Party: Principal Investigator, Dianne Bryant, Associate Professor, University of Western Ontario, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FKSMC 2010 - 4
Record Dates: First submitted 2012-06-04; First posted 2012-06-15 (Estimated); Last update posted 2014-04-25 (Estimated); Status verified 2014-04

CONDITIONS: Bankart Lesions; Anterior Shoulder Instability
Keywords: Shoulder; Bankart; Anterior Instability; Rotator Cuff
MeSH Terms: conditions — Bankart Lesions

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arthroscopic Bankart Repair & Rotator Interval Closure (Active Comparator)
  Interventions: Procedure: Closure of rotator interval
- Arthoscopic Bankart Repair alone (Active Comparator)
  Interventions: Other: Arthroscopic Bankart Repair alone

INTERVENTIONS:
Other: Arthroscopic Bankart Repair alone — Usual arthroscopic Bankart repair
  Arms: Arthoscopic Bankart Repair alone
Procedure: Closure of rotator interval — Usual arthroscopic Bankart repair plus rotator cuff interval closure
  Arms: Arthroscopic Bankart Repair & Rotator Interval Closure

SUMMARY:
The null hypothesis is that there is no statistical difference between the two treatment groups for any outcome. The investigators suspect that patients who undergo a Bankart lesion repair with rotator interval closure will have lower quality of life and less external rotation compared to patients who undergo a Bankart lesion repair alone. No difference will be observed for recurrence rate between the two treatment groups

DETAILED DESCRIPTION:
Research assessing the role and effectiveness of rotator interval closure is important to attempt to determine the most beneficial and efficient treatment for Bankart lesions and anterior shoulder instability. To date there is only weak evidence supporting the superiority of Bankart lesion repair in addition to rotator interval closure compared to Bankart lesion repair alone.

Does Bankart lesion repair with rotator interval closure result in differences in quality of life, range of motion and recurrence at 3 weeks, 6 weeks, 3 months, 6 months, 1 year and 2 years in similar patients with Bankart lesions who are treated with Bankart lesion repair alone?

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 15 to 50 years
* At least one episode of demonstrated dislocation
* Bankart lesion of the anterior glenoid labrum
* Absence of other capsular and tendon injuries
* Absence of glenoid fractures or divots

Exclusion Criteria:

* Posterior instability or the need for posterior surgical reconstruction
* Significant bone lesions greater than 3mm of the humeral head anterior-to- posterior (Hill-Sachs lesions)
* Presence of other pathologic conditions of the shoulder (excluding SLAP lesions)

Ages: 15 Years to 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 142 (Estimated)
Dates: Start 2010-02; Primary Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
Western Ontario Shoulder Instability Index | 3,6 weeks;3,6 months; 1,2 years
  Disease-specific quality of life measurement tool (21 questions, 4 domains)

SECONDARY OUTCOMES:
Range of Motion | 3,6 months; 1-2 years
  * Universal goniometer
  * Internal & external ROM at neutral (0°) and 90° of abduction
  * Both active and passive ROM at both positions
4-Item Pain Intensity Measure | 3,6, weeks; 3, 6 months; 1,2 years
  Pain intensity in the morning, afternoon, evening and with activity
Upper Extremity Functional Index | 3,6 weeks; 3,6 months; 1,2 years
  Limb-specific quality of life measurement tool (20 questions)
Recurrence | 3,6 weeks; 3,6 months; 1,2 years
  Patient-reported re-dislocation

CONTACTS AND LOCATIONS:
Overall Officials: Dianne Bryant, PhD, Study Director — The University of Western Ontario
Locations (1):
- London Health Sciences Centre - Unviersity Hospital, London, Ontario, Canada